CLINICAL TRIAL: NCT02512224
Title: Comparison of Short-term Mortality and Morbidity Between Parenteral and Enteral Nutrition for Adults Without Cancer: a Propensity-matched Analysis Using a National Inpatient Database
Brief Title: Comparison of Outcomes Between Parenteral and Enteral Nutrition
Status: Completed | Type: Observational
Sponsor: Tokyo University (Other)
Responsible Party: Principal Investigator, Sumito Ogawa, Associate Professor, Tokyo University
Other Study IDs: MHLW H26-Policy-011; MHLW H26-Special-047 (Other Grant/Funding Number: Ministry of Health, Labour and Welfare, Japan); NCGG 25-11 (Other Grant/Funding Number: National Center for Geriatrics and Gerontology , Japan)
Record Dates: First submitted 2015-07-28; First posted 2015-07-30 (Estimated); Results first posted 2015-09-10 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Deglutition Disorders
Keywords: parenteral nutrition; enteral nutrition
MeSH Terms: conditions — Deglutition Disorders; Hyperphagia | interventions — Parenteral Nutrition; Enteral Nutrition

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parenteral nutrition: investigators selected participants aged 20 years or older who had undergoneparenteral nutrition by central venous port insertion between April 1, 2012, and March 31, 2013.
  Interventions: Device: Parenteral nutrition
- Enteral nutrition: investigators selected participants aged 20 years or older who had undergone enteral nutrition by percutaneous endoscopic gastrostomy, percutaneous transesophageal gastrotubing, or ileostomy between April 1, 2012, and March 31, 2013.
  Interventions: Device: Enteral nutrition

INTERVENTIONS:
Device: Parenteral nutrition — Participants are retrospectively selected with propensity score matching
  Groups: Parenteral nutrition
Device: Enteral nutrition — Participants are retrospectively selected with propensity score matching
  Groups: Enteral nutrition

SUMMARY:
Short-term outcomes of parenteral and enteral nutrition for patients unable to eat normally were compared and analyzed.

DETAILED DESCRIPTION:
Data were acquired from patients selected from a national inpatient database covering 1,057 hospitals in Japan. Participants had received artificial nutrition between April 2012 and March 2013, were 20 years or older, and did not have cancer. Participants were grouped into two groups: those receiving parenteral nutrition and those receiving enteral nutrition. The investigators performed one-to-one propensity-score matching between the groups. The primary outcome measurements were mortality rates at 30 and 90 days after the start of the procedure. The secondary outcomes were post-procedural complications, pneumonia, and sepsis. The investigators analyzed survival length of stay after the procedure using a Cox proportional hazards model.

ELIGIBILITY:
Inclusion Criteria:

* investigators selected participants aged 20 years or older who had undergone either parenteral nutrition by central venous port insertion or enteral nutrition by percutaneous endoscopic gastrostomy, percutaneous transesophageal gastrotubing, or ileostomy between April 1, 2012, and March 31, 2013. Patients who received both gastrostomy and central venous port insertion were assigned to the gastrostomy group.

Exclusion Criteria:

* investigators excluded participants who had been diagnosed with cancer.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this study, the investigators used the Japanese Diagnosis Procedure Combination database, the details of which have been described elsewhere. The database includes administrative claims and discharge abstract data. In 2012, these data were collected for about seven million inpatients from 1,057 participating hospitals across Japan, which amounted to about half of the acute-care hospitalizations in the country.
Sampling Method: Non-Probability Sample
Enrollment: 5824 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumito Ogawa, MD. PhD., Principal Investigator — Tokyo University

REFERENCES:
- [Derived] Tamiya H, Yasunaga H, Matusi H, Fushimi K, Akishita M, Ogawa S. Comparison of short-term mortality and morbidity between parenteral and enteral nutrition for adults without cancer: a propensity-matched analysis using a national inpatient database. Am J Clin Nutr. 2015 Nov;102(5):1222-8. doi: 10.3945/ajcn.115.111831. Epub 2015 Oct 7. PMID 26447149

RESULTS

PARTICIPANT FLOW:
Groups:
- Parenteral Nutrition: investigators selected participants aged 20 years or older who had undergoneparenteral nutrition by central venous port insertion between April 1, 2012, and March 31, 2013.
  Parenteral nutrition and Enteral nutrition: Participants are retrospectively selected with propensity score matching
- Enteral Nutrition: investigators selected participants aged 20 years or older who had undergone enteral nutrition by percutaneous endoscopic gastrostomy, percutaneous transesophageal gastrotubing, or ileostomy between April 1, 2012, and March 31, 2013.
  Parenteral nutrition and Enteral nutrition: Participants are retrospectively selected with propensity score matching
Period: Overall Study
Arm/Group | Parenteral Nutrition | Enteral Nutrition
Started | 2912 | 2912
Completed | 2912 | 2912
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parenteral Nutrition | Enteral Nutrition | Total
Number analyzed (Participants) | 2912 | 2912 | 5824
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 390 | 354 | 744
  >=65 years | 2522 | 2558 | 5080
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.43 (14.086) | 78.81 (13.558) | 78.62 (13.824)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1460 | 1437 | 2897
  Male | 1452 | 1475 | 2927
Region of Enrollment [Number; unit: participants]
  Japan | 2912 | 2912 | 5824

OUTCOME MEASURES:

1. Primary Outcome: Mortality Calculated From Outcome Section From DPC Database at 90 Days
Time Frame: 90 days after the start of the procedure
Measure: Number; unit: Participants
Arm/Group | Parenteral Nutrition | Enteral Nutrition
Number analyzed (Participants) | 2912 | 2912
Participants | 359 | 287

2. Secondary Outcome: Post-procedural Pneumonia
Time Frame: the incidence of post-procedural pneumonia occurring during hospitalization. Participants will be followed for the duration of hospital stay, an expected median of 3 weeks after procedure.
Measure: Number; unit: Participants
Arm/Group | Parenteral Nutrition | Enteral Nutrition
Number analyzed (Participants) | 2912 | 2912
Participants | 346 | 450

3. Secondary Outcome: Post-procedural Sepsis
Time Frame: the incidence of post-procedural sepsis occurring during hospitalization. Participants will be followed for the duration of hospital stay, an expected median of 3 weeks after procedure.
Measure: Number; unit: Participants
Arm/Group | Parenteral Nutrition | Enteral Nutrition
Number analyzed (Participants) | 2912 | 2912
Participants | 129 | 108

4. Secondary Outcome: Re-admission 30 Days
Time Frame: re-admission within 30 days of discharge.
Measure: Number; unit: Participants
Arm/Group | Parenteral Nutrition | Enteral Nutrition
Number analyzed (Participants) | 2912 | 2912
Participants | 188 | 159

5. Secondary Outcome: Mortality Calculated From Outcome Section From DPC Database at 14 Days
Time Frame: 14 days after the start of the procedure
Measure: Number; unit: Participants
Arm/Group | Parenteral Nutrition | Enteral Nutrition
Number analyzed (Participants) | 2912 | 2912
Participants | 114 | 89

6. Secondary Outcome: Mortality Calculated From Outcome Section From DPC Database at 30 Days
Time Frame: 30 days after the start of the procedure
Measure: Number; unit: participants
Arm/Group | Parenteral Nutrition | Enteral Nutrition
Number analyzed (Participants) | 2912 | 2912
participants | 114 | 89

ADVERSE EVENTS:
Arm/Group | Parenteral Nutrition | Enteral Nutrition
Serious Adverse Events (participants affected / at risk) | 0/2912 | 0/2912
Other Adverse Events (participants affected / at risk) | 0/2912 | 0/2912

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No